CLINICAL TRIAL: NCT04412044
Title: Effect of Anti-interleukin 5 (IL5) Therapy on Sputum Cells and Cytokines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Tatjana Decaesteker, Principal Investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s58608
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Asthmatics (Experimental): Patients receive anti-IL5 treatment as part of their prescribed routine. Immunological and clinical parameters will be evaluated at the start of the treatment and after 6 months of treatment
  Interventions: Drug: Mepolizumab Injection [Nucala]

INTERVENTIONS:
Drug: Mepolizumab Injection [Nucala] — Patients receive monthly injection with 100 mg mepolizumab
  Other Names: Anti-IL5 treatment

SUMMARY:
22 asthmatics, in which mepolizumab was to be started, gave permission for inclusion and were followed up prospectively. Clinical and lung functional data, sputum analyses and cytokine measurements were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 < 80% in the last 12 months
* use of high dose inhaled corticosteroids (ICS) in combination with other additional medication or continuous use of oral corticosteroids (OCS)
* at least 2 exacerbations in the last 12 months
* at least 300 blood eosinophils/µl once in the last 12 months and at the time of inclusion
* Anti-IL5 treatment prescribed by the physician

Exclusion Criteria:

* Not completing all visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Airway inflammation | Day 1 and after 6 months
  Bronchial airway inflammation. Differential cell count will be performed on sputum samples, determining eosinophilic (>3% eosinophils, <61% neutrophils), neutrophilic (<3% eosinophils and >61% neutrophils), pauci-granulocytic (<3% eosinophils and <61% neutrophils) and mixed granulocytic airway inflammation (>3% eosinophils and >61% neutrophils).
Change in Forced Expiratory Volume in 1 seconds (FEV1) | Day 1 and after 6 months
  The forced expiratory Volume in 1 second will be measured using spirometry

SECONDARY OUTCOMES:
Cytokine pattern in the airways | Day 1 and after 6 months
  Cytokines concentrations (pg/ml) will also be determined in sputum supernatant using a U-plex assay.
Cytokine pattern in the bloodstream | Day 1 and after 6 months
  Cytokines concentrations (pg/ml) will also be determined in serum using a U-plex assay.
Change in asthma control | Day 1 and after 6 months
  Asthma control will be determined using the Asthma Control Questionnaire (ACQ-6), including 6 questions. Each question will be scored from 0-6 and added together. This final score will be divided by the number of questions. If ACQ-6 < 0.75 = controlled asthma, ACQ-6 from 0.75-1.5 = partly controlled asthma and ACQ-6 > 1.5 = uncontrolled asthma.
Biomarkers for airway inflammation | Day 1 and after 6 months
  Fraction exhaled Nitric Oxid (FeNO) will be used as biomarker for eosinophilic airway inflammation. FeNO < 25 ppb = eosinophilic inflammation less likely, FeNO between 25 and 50 ppm = need further interpretation with additional clinical information, FeNO > 50 ppm = indication of eosinophilic airway inflammation (according to the American Thoracic Society guidelines)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Decaesteker, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: No